CLINICAL TRIAL: NCT00514072
Title: A Double-Blind Randomized Phase 2.5 Trial of ONY-P1 Vaccine Versus Placebo in Men With D0 Prostate Cancer Following Limited Androgen Ablation
Brief Title: Vaccine Therapy in Treating Patients With Stage D0 Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kael-GemVax Co., Ltd. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000559937; NCI-07-C-0188; ONYVAX-ONY-P1-07-01
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Experimental): Patients receive ONY-P1 vaccine with BCG intradermally on days 1 and 15. Patients then receive ONY-P1 vaccine alone on day 29 and then every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: BCG vaccine; Biological: prostate cancer vaccine ONY-P1
- Arm II (Placebo Comparator): Patients receive placebo vaccine intradermally on days 1, 15, and 29 and then every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: BCG vaccine — given intradermally
  Arms: Arm I
Biological: prostate cancer vaccine ONY-P1 — given intradermally
  Arms: Arm I
Other: placebo — given intradermally
  Arms: Arm II

SUMMARY:
RATIONALE: Vaccines made from tumor cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This randomized phase II trial is studying vaccine therapy to see how well it works compared with a placebo in treating patients with stage D0 prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether ONY-P1 vaccine can increase the time to PSA-defined progression in patients with androgen-dependent stage D0 prostate cancer.

Secondary

* To evaluate all toxicities related to ONY-P1 vaccine.
* To compare the immunologic response in patients treated with ONY-P1 vaccine vs placebo.
* To evaluate PSA kinetics (doubling time/velocity) of treatment.
* To evaluate time to testosterone recovery following limited androgen ablation.

OUTLINE: Patients are stratified according to estimated PSA doubling time (< 12 months vs ≥ 12 months).

Patients receive goserelin subcutaneously once. Approximately 3 months later, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive ONY-P1 vaccine with BCG intradermally on days 1 and 15. Patients then receive ONY-P1 vaccine alone on day 29 and then every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive placebo vaccine intradermally on days 1, 15, and 29 and then every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 15 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathological documentation of prostate cancer

  * If no pathologic specimen is available, patients may enroll on study with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease
* Biochemical progression, as defined by the following:

  * A rise in PSA of ≥ 2 ng/mL above the nadir (for patients previously treated with definitive radiotherapy or cryotherapy)
  * Two consecutive rises in PSA > 0.3 ng/mL (for patients previously treated with radical prostatectomy)
* PSA ≤ 20 ng/mL
* Testosterone ≥ lower limit of normal
* Negative CT scan and bone scan for metastatic prostate cancer
* No clinically active brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-1
* Life expectancy ≥ 6 months
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 1.5 mg/dL OR total bilirubin ≤ 3.0 mg/dL (in patients with Gilbert's syndrome)
* AST and ALT ≤ 2.5 times upper limit of normal
* No other active malignancies within the past 60 months (with the exception of nonmelanoma skin cancer or carcinoma in situ of the bladder)
* No life-threatening illnesses
* No immunocompromised status due to any of the following:

  * HIV positivity
  * Active autoimmune diseases, such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjögren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome, or active Grave's disease

    * Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function, including CNS, heart, lungs, kidneys, skin, or gastrointestinal tract, will be allowed
  * Other immunodeficiency diseases or iatrogenic immunodeficiency from drugs
* No other serious medical illness that would interfere with the patient's ability to carry out the treatment program
* No documented contraindication (allergy or severe reaction to BCG)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy, including surgery and radiotherapy (no toxicity ≥ grade 2)
* No prior chemotherapy
* No concurrent topical steroids (including steroid eye drops) or systemic steroids

  * Nasal or inhaled steroid use is permitted
* No concurrent medications used for urinary symptoms, including 5-alpha reductase inhibitors (finasteride and dutasteride)
* No concurrent alternative medications known to alter PSA (e.g., phytoestrogens or saw palmetto)
* No other concurrent hormonal therapy
* No other concurrent anticancer treatment, including chemotherapy, systemic glucocorticoids, radiotherapy, major surgical procedures for prostate cancer, or nonprotocol-related immunotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-03; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Time to PSA progression

SECONDARY OUTCOMES:
Toxicity
Immunologic response as assessed by ELISPOT assay
PSA kinetics (doubling time/velocity) of treatment
Time to testosterone recovery

CONTACTS AND LOCATIONS:
Overall Officials: James L. Gulley, MD, PhD, FACP, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aragon-Ching JB, Williams KM, Gulley JL. Impact of androgen-deprivation therapy on the immune system: implications for combination therapy of prostate cancer. Front Biosci. 2007 Sep 1;12:4957-71. doi: 10.2741/2441. PMID 17569623
- [Derived] Huang J, Jochems C, Talaie T, Anderson A, Jales A, Tsang KY, Madan RA, Gulley JL, Schlom J. Elevated serum soluble CD40 ligand in cancer patients may play an immunosuppressive role. Blood. 2012 Oct 11;120(15):3030-8. doi: 10.1182/blood-2012-05-427799. Epub 2012 Aug 28. PMID 22932804